CLINICAL TRIAL: NCT05052476
Title: First Line Dose-efficacy Study of Bactecal® D Liquid for Infant Colic
Acronym: BACTECOLIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Astel Medica (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BACTECOLIC
Record Dates: First submitted 2021-09-09; First posted 2021-09-22 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-07

CONDITIONS: Colic
MeSH Terms: conditions — Colic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Open label Bactecal® D Liquid 1 dose (Experimental): Patients will receive 1 dose of Bactecal® D Liquid by day which corresponds to 2 ml of product
  Interventions: Dietary Supplement: Bactecal® D Liquid
- Open label Bactecal® D Liquid 2 doses (Experimental): Patients will receive 2 doses of Bactecal® D Liquid by day which correspond to 4 ml of product.
  Interventions: Dietary Supplement: Bactecal® D Liquid

INTERVENTIONS:
Dietary Supplement: Bactecal® D Liquid — The patients will be randomized into two arms, A and B, in function of the intervention dose

SUMMARY:
This randomized, open label, dose-response study will be realized at the first line with Bactecal® D Liquid. The objective is to investigate Bactecal® D Liquid in the context of infantile colics.

The patients will be randomized into two arms, A and B, in function of the intervention dose. The quality of life of te parents as well as the daily median crying time and the number of daily crying will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Full term healthy infant (37-41 weeks amenorrhea)
* Birth weight >2750 g
* Aged between 2 and 8 weeks
* Presenting symptoms of infant colic as defined by Rome IV criteria by Zeevenhoven et al. 2017
* Signed written informed consent of the parent/tutor

Exclusion Criteria:

* Premature birth
* Using probiotics as a treatment, different from the one that could contain the formula at the time of study recruitment
* Acute or chronic illness as judged by the investigator which avoids the participation to the study .
* Parents unable to understand the requirements of study participation as judged by the investigator
* Malnutrition as judged by a body weight/height ratio <5 %

Ages: 2 Weeks to 8 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 68 (Actual)
Dates: Start 2022-04-08 (Actual); Primary Completion 2023-10-08 (Actual); Study Completion 2023-10-16 (Actual)

PRIMARY OUTCOMES:
Change in parent quality of life (QoL) score | Change from baseline parent QoL score at 28 days
  By measuring parent quality of Life (QoL) score. Scale from 1 (minimum) to 7 (maximum). Higher scores mean a better outcome.

SECONDARY OUTCOMES:
Change of daily median crying time | Change from baseline daily median crying time at 28 days
  By measuring the mean change in crying time
Change of the number of crying | Change from baseline number of crying at 28 days
  By measuring the numbers per day

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Brussel, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No